CLINICAL TRIAL: NCT06939699
Title: The Effect of Social Media-Based Education on Women's Knowledge, Attitudes, and Health Literacy Regarding Cancer Screenings: A Randomized Controlled Trial
Brief Title: Social Media-Based Education on Cancer Screening Awareness in Women: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Ergin (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor-Investigator, Emine Ergin, Associate professor, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBU-SC2025-RCT
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer Screening; Breast Cancer Screening; Colorectal Cancer Screening; Digital Health Literacy
Keywords: internet based intervention; cancer screening; social media; health literacy; education

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: the social media-based education group or the standard online education group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Media-Based Education Group (Experimental): Participants in this group will receive daily infographic/video-based education for 8 weeks via WhatsApp or Instagram. The content focuses on cancer screening awareness (breast, cervical, colorectal) and digital health literacy. The educational content is developed based on the Socio-Ecological Model.
  Interventions: Behavioral: Social Media-Based Education
- Standard Education Group (Active Comparator): Participants in this group will receive two standard 40-minute online educational sessions using PowerPoint presentations via Microsoft Teams/Zoom, one week apart. Content includes cancer screening and digital health literacy information.
  Interventions: Behavioral: Standard Online Education

INTERVENTIONS:
Behavioral: Social Media-Based Education — This intervention includes daily delivery of 56 infographic/video-based educational materials over 8 weeks via WhatsApp or Instagram. The content focuses on awareness of breast, cervical, and colorectal cancer screenings, healthy lifestyle behaviors, and digital health literacy. The materials are developed based on the Socio-Ecological Model.
  Other Names: Instagram & WhatsApp Infographic Education
  Arms: Social Media-Based Education Group
Behavioral: Standard Online Education — Participants receive two 40-minute online educational sessions one week apart via Microsoft Teams/Zoom. The content includes cancer screening awareness (breast, cervical, colorectal), preventive strategies, and the use of digital health tools such as e-Nabız and MHRS.
  Arms: Standard Education Group

SUMMARY:
This randomized controlled trial investigates the impact of a social media-based educational program on women's knowledge, attitudes, and digital health literacy regarding breast, cervical, and colorectal cancer screenings. The intervention is based on the Socio-Ecological Model and aims to improve awareness and screening participation. Participants in the intervention group receive daily educational content for 8 weeks via social media platforms (WhatsApp/Instagram), while the control group receives two standard online education sessions via Microsoft Teams app. The study includes 132 women aged 30 to 70 in Türkiye who have not previously participated in cancer screenings. The primary outcomes include changes in cancer knowledge, attitudes, and digital health literacy levels measured by validated scales.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to evaluate the effect of a social media-based educational intervention on women's knowledge, attitudes, and digital health literacy regarding cancer screenings. The trial will include 132 women between the ages of 30 and 70 who have never undergone breast, cervical, or colorectal cancer screening. Participants are recruited through health institutions and randomized into two parallel groups: the intervention group and the control group.

The educational intervention was developed in accordance with the Socio-Ecological Model (SEM), incorporating individual, interpersonal, institutional, community, and policy-level messages. The intervention group receives 56 infographics and/or videos total over 8 weeks via closed WhatsApp and Instagram groups. The content includes evidence-based information on cancer epidemiology, risk factors, symptoms, screening methods, healthy lifestyle behaviors, and digital health tools such as e-Nabız and MHRS.

The control group receives traditional education via two 40-minute online sessions (1 week apart), covering the same content without daily engagement. The outcomes will be measured using validated instruments to assess changes in participants' knowledge of cancer screenings, their attitudes towards screening, and their digital health literacy. Data collection will take place before and after the intervention period. The study has been approved by the Istanbul Medipol University Non-Interventional Clinical Research Ethics Committee (Approval Number: E-10840098-202.3.02-7880).

This research is expected to contribute to public health strategies that use digital platforms to enhance cancer screening behaviors and improve health literacy among women.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 30 to 70 years
* Use Instagram and/or WhatsApp actively
* Literate and able to complete online forms
* Voluntarily consent to participate

Exclusion Criteria:

* Diagnosed with any type of cancer
* Have undergone previous cancer screening

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Change in Cancer Screening Knowledge Score | Baseline and 4 weeks after the intervention
  Measured using a validated cancer screening knowledge questionnaire. Total score reflects level of knowledge about breast, cervical, and colorectal cancer screening guidelines.
Change in Attitudes Toward Cancer Screening | Baseline and 4 weeks after the intervention
  Assessed using a Likert-type scale measuring women's attitudes toward cancer screening behavior and participation.
Change in Digital Health Literacy Level | Baseline and 4 weeks after the intervention
  Evaluated using the eHealth Literacy Scale adapted to Turkish. Assesses ability to search, understand, and apply online health information.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Çınar, phD candidate midwife, Study Chair — Health Science University
Locations (1):
- Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study involves sensitive data based on personal health information and is conducted with a limited number of participants as part of a doctoral thesis. Therefore, there is no plan to share individual participant data (IPD) directly with other researchers.